CLINICAL TRIAL: NCT01610258
Title: Contribution of the Study of Maternal Plasmatic Regulator T Cells and Th17 for the Diagnosis of Acute Chorioanmionitis Among Women Hospitalized for Premature Rupture of Fetal Membranes (PPROM) Between 24 and 34 Gestation Weeks
Brief Title: Maternal Plasmatic Regulatory T Cells and Th17 as Possible Diagnosis Markers of Acute Chorioamnionitis
Acronym: ICAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BARDOU-PHRC-2011
Record Dates: First submitted 2012-05-31; First posted 2012-06-01 (Estimated); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Pathology of Pregnancy
Keywords: pregnancy, chorioamnionitis, PPROM, Treg
MeSH Terms: conditions — Chorioamnionitis; Preterm Premature Rupture of the Membranes | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Blood and placenta samples — The placenta sample is realised, specially for the study, in surgical unit after the delivery.
  The blood samples are taken, specially for the study, the day of admission and at time of delivery or seven days after the admission.

SUMMARY:
The purpose of this study is to evaluate if regulator T cells (Treg) and Th17 level modifications in maternal blood and placenta could be correlated to a chorioamnionitis, in women hospitalized for PPROM.

DETAILED DESCRIPTION:
Acute chorioamnionitis is the principal antecedent of premature birth and an important contributor to specific neonatal and other complications that may extend throughout subsequent life. The PPROM is a high risk condition for developing chorioamnionitis. Available biological markers have a low prognostic value. Indeed, currently the diagnosis of intra-uterine infection relies only on placental cultures and anatomo-pathological exam after the delivery.

Moreover, pregnancy is an immunologic particular condition. Indeed an immune tolerance is required with respect to the fetus and is mediated by Treg lymphocytes, which suppressed Th17 activity.

Recent studies have shown among women with frequent miscarriages, a balance between Treg and Th17, with a decrease in Treg number and an increase in Th17 number in decidua and blood.

In case of infection, the immune pro-inflammatory response (Th17) is restored in peripheric tissues and in blood in order to limit the extention of intra-uterine infection. This restoration of this pro-inflammatory response could be due to a modification of Treg number ou tolerogenic activity.

In this context, our hypothesis is that chorioamnionitis will lead to a decrease of treg proportion and an increase of Th17 proportion in lymphocyte populations of maternal blood and placenta, with a back to values near than which is observed in beginning of pregnancy or in no pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed
* Patient affiliated with a social security scheme
* term pregnancy betwwen 24 and 34 weeks
* PPROM diagnosis
* singleton pregnancy

Exclusion Criteria:

* delivery occured in 1 hour after admission
* hemorragic praevia placenta or retro-placental hematoma
* confirmed autoimmune or inflammatory disease
* confirmed infectious disease by VIH, VHC, and VHB

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2013-03-26 (Actual); Primary Completion 2016-12-08 (Actual); Study Completion 2016-12-08 (Actual)

PRIMARY OUTCOMES:
Evaluate the percentage of Treg in maternal blood at the time of admission | the day of delivery or 7 days after the admission if no delivery

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Maternité du CHU de Dijon, Dijon, Bourgogne-Franche-Comté
  - Hôpital Hautepierre, Strasbourg